CLINICAL TRIAL: NCT01018108
Title: Effect of Acupuncture on Brain Serotonin Among Breast Cancer Survivors
Brief Title: Visualization of the Effect of Acupuncture on Brain Serotonin in Breast Cancer Survivors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCC 17108
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Photons; Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Other): Patients undergo acupuncture twice weekly for 2 weeks and then once weekly for 6 weeks. Patients undergo single photon emission computed tomography imaging with iodine 123-I ADAM before and after completion of acupuncture.
  Interventions: Procedure: Single Photon Emission Computed Tomography; Procedure: Acupuncture Therapy; Other: Questionnaire Administration; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Single Photon Emission Computed Tomography — Undergo single photon emission computed tomographt imaging
  Other Names: SPECT imaging, tomography, emission computed, single photon
Procedure: Acupuncture Therapy — Undergo acupuncture
  Other Names: Acupuncture
Other: Questionnaire Administration — Ancillary study
Other: Laboratory Biomarker Analysis — Correlative Study

SUMMARY:
RATIONALE: New imaging procedures, such as single photon emission computed tomography, may help in learning how acupuncture affects serotonin levels in the brain of breast cancer survivors. PURPOSE: This phase I trial is studying the best way to visualize the effect of acupuncture on brain serotonin in breast cancer survivors.

DETAILED DESCRIPTION:
Detailed Description

OBJECTIVES:

I. To determine the feasibility of using [123-I] ADAM Serotonin transporter (SERT) binding as a putative biomarker to visualize the mechanism of effects of acupuncture for hot flashes involving serotonin.

OUTLINE: Patients undergo acupuncture twice weekly for 2 weeks and then once weekly for 6 weeks. Patients undergo single photon emission computed tomography imaging with iodine 123-I ADAM before and after completion of acupuncture.

After completion of study treatment, patients are followed for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* History of Stage I, II, or III breast cancer for at least 12 months
* Have been seen by an oncologist within the previous 6-month period and determined to be free of disease by clinical examination and history
* Have been receiving endocrine therapy (tamoxifen or aromatase inhibitors for at least four weeks)
* Experienced hot flashes with a hot flash composite score of 5 or greater per day
* Hot flashes have been present for at least a month before study entry

Exclusion Criteria:

* Currently on chemotherapy or radiation therapy as adjuvant treatment
* Started with hormonal therapies such as tamoxifen or aromatase inhibitors within the last 4 weeks; or plan to change or terminate hormonal therapies in the next 14 weeks
* Any history of use of psychotropic medication such as SSRI use for the past 6 months
* Any past use of centrally acting medications such as clonidine for the past 6 months
* Any past diagnosis of a Major Depressive Episode within the last 6 months
* Any allergy to iodine or shell-fish or radio-nuclear materials
* Current use of estrogen and/or progestin
* Pregnancy
* Breast feeding
* Women of child-bearing potential NOT willing to use a medically acceptable form of contraception
* Current use of any anti-convulsant such as gabapentin
* History of cerebral infarction (including lacunar infarct with symptoms >= 24 hours duration)
* History of Binswanger's disease (or a history of hypertensive encephalopathy)
* History of intracranial hemorrhage
* History of head trauma with loss of consciousness
* History of encephalitis
* History of extended exposure to known neurotoxin (e.g., cyanide, carbon monoxide)
* Uncontrolled metabolic disorder (e.g., thyroid disease, diabetes mellitus)
* History of normal pressure hydrocephalus
* History of Parkinson's or other basal ganglia disease
* History of substance abuse in the previous 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
SERT uptake ratios
Hot flash composite score (HFCS)

SECONDARY OUTCOMES:
Hot flash related daily interference scale (HFRDIS)
Pittsburgh sleep quality index (PSQI)
Brief Fatigue Inventory (BFI)
HADS
Global assessment scale
Hot flash frequency and severity
Acupuncture expectancy scale
Credibility rating of acupuncture

CONTACTS AND LOCATIONS:
Overall Officials: Jun Mao, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States